CLINICAL TRIAL: NCT06800170
Title: Treatment of Menstrual Cycle Alterations in Adolescents
Acronym: HP-phD_Adolesc
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Principal Investigator, Vittorio Unfer, Professor, AGUNCO Obstetrics and Gynecology Centre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP+phD in adolescents
Record Dates: First submitted 2025-01-16; First posted 2025-01-29 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-07

CONDITIONS: Amenorrhea; Oligomenorrhea; PCOS (Polycystic Ovary Syndrome)
Keywords: myo-Inositol; Dioscorea Villosa; adolescents
MeSH Terms: conditions — Amenorrhea; Oligomenorrhea; Polycystic Ovary Syndrome | interventions — Inositol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated Group HP+phD (Experimental)
  Interventions: Dietary Supplement: myo-Inositol plus DIoscorea Villosa
- Controls (No Intervention): Not treated patients

INTERVENTIONS:
Dietary Supplement: myo-Inositol plus DIoscorea Villosa — myo-Inositol + alpha-lactalbumin + folic acid once daily, Dioscorea Villosa + alpha-lactalbumin + Vitamin D twice daily
  Other Names: myo-Inositol; Dioscorea Villosa
  Arms: Treated Group HP+phD

SUMMARY:
the aim of the present study is intended to evaluate how treatment with Myo-Inositol and Dioscorea Villosa can help improve menstrual cycle irregularities in adolescents, both with and without PCOS.

DETAILED DESCRIPTION:
The present study aims to evaluate the possible beneficial effect of a treatment with Inofolic HP combined with Inofolic phD on the improvement if menstrual cycle alteration in adolescent patients with or without PCOS.

The molecules chosen for the study are the following: myo-Inositol, α-lactalbumin, Dioscorea Villosa, and Vitamin D, are already commercialized as dietary supplements, commonly administered at same dosage provided in the present study, also for prolonged treatments, with no side effects associated.

ELIGIBILITY:
Inclusion Criteria:

* adolescent women aged 14-19 years old, with at least 3 years passed after menarche, and oligomenorrhea or amenorrhea

Exclusion Criteria:

* Primary amenorrhea.
* Hyperandrogenism due to other factors (i.e. adrenal hyperplasia or Cushing syndrome).
* Hyperprolactinemia or overt hypothyroidism (TSH ≥4).
* Other hormonal alterations.
* Ongoing hormonal therapies, including OCPs, six months before enrollment.
* Ongoing pharmacological therapies.
* Ongoing use of myo-Inositol supplement or other source of myo-Inositol, or Dioscorea villosa, six months before enrollment.

Ages: 14 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Female patients
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Menstrual cycle regularity | 6 months
  The intervention is targed to adolescent patients suffering from menstrual cycle alterations. Particularly, we aim to asses the regularization of the menstrual cycle in those patients with polimenhorrea and oligo-/ amenorrhea, with irregular menstrual cycle (shorter than 21 days or longer than 35 days).
  The purpose of the study is to compare the percentage of patients exhibiting a regular menstrual cycle at the end of the treatment period, in the study group vs control.

CONTACTS AND LOCATIONS:
Locations (3):
- Zhordania and Khomasuridze Institute of Reproductology, Tbilisi, Georgia, Georgia
- Agunco, Rome, Italy, Italy
- Department of Obstetrics and Gynecology with Reproductive Medicine, F.I. Inozemtsev Academy of Medical Education, Saint Petersburg, Russian Federation, Russia

IPD SHARING:
Plan to Share IPD: No